CLINICAL TRIAL: NCT00269009
Title: CHERL, Connecting Primary Care Patients With Community Resources to Facilitate Behavior Change
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Great Lakes Research Into Practice Network (Network)
Collaborators: Robert Wood Johnson Foundation (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Michigan Department of Community Health (Other); Marquette General Health System (Other); Upper Peninsula Health Education Corporation; (Unknown); Grand Rapids Medical Education and Research Center for Health Professions (Other); Greater Flint Health Coalition (Other); Genesee Health Plan (Unknown); Genesys Health System (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: 61-9165
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2006-09

CONDITIONS: Tobacco Use Disorder; Alcohol Abuse; Lack of Physical Activity; Poor Diet
Keywords: Tobacco use
MeSH Terms: conditions — Tobacco Use Disorder; Alcoholism; Sedentary Behavior; Tobacco Use

INTERVENTIONS:
Behavioral: CHERL

SUMMARY:
The investigators want to find out if providing a Community Health Educator Referral Liaison (CHERL) helps practices help their patients change risky behaviors (tobacco use, physical inactivity, unhealthy diet, and risky drinking) by connecting patients to available services in the community or directly providing behavior change support.

DETAILED DESCRIPTION:
What is this about? Prescription for Health (P4H) is a national initiative funded by the Robert Wood Johnson Foundation. Nine projects have been funded nationally in this second round to advance the goals of improving health behavior identification and delivery in primary care practice. Each project is conducted through a practice-based research network (PBRN). In Michigan, our PBRN is called the Great Lakes Research In Practice Network (GRIN).

What is the purpose of the CHERL project? In our study, we want to find out if providing a Community Health Educator Referral Liaison (CHERL) helps practices help their patients change risky behaviors (tobacco use, physical inactivity, unhealthy diet, and risky drinking) by connecting patients to available services in the community or directly providing behavior change support.

Primary care providers play a key roll in encouraging patients to choose healthy behaviors. However, effective behavior change requires long term follow up and support that may not be readily available within the office practice. CHERL can help provide or link to those services thus helping the healthy message promoted by the clinician to have a more powerful and lasting effect.

What is the CHERL intervention? With this funding, we will hire and train a CHERL to work with practices. The purpose of the CHERL is for him/her to help secure behavior change support for your patients either by referring to an available resource within the community or directly providing the service. This service is available to patients with or without chronic disease diagnoses (i.e, patients with diabetes, heart disease, hypertension, obesity, back pain, lung disease, or generally healthy with opportunities to change unhealthy habits).

Patients are referred to the CHERL and he/she will determine an appropriate next step for your patient - either referral to a community program or the CHERL will provide brief telephone counseling. The health care provider will receive feedback specifically on each patient referred.

In addition, some practices (consultant-enhanced) will receive additional assistance from the CHERL, as he/she serves as a consultant to the practice, helping the practice to identify systematic mechanisms for identification and referral of at risk patients to the CHERL.

ELIGIBILITY:
Inclusion Criteria:

* Patients, clinicians, and their staff participating in this GRIN study.

Exclusion Criteria:

* Patients, clinicians, and their staff who are not participating in this GRIN study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-01; Study Completion 2007-02

PRIMARY OUTCOMES:
The primary outcome of interest is the referral rate for any unhealthy behavior to the CHERL with the predictor variable being referral-only versus consultant-enhanced practices.

SECONDARY OUTCOMES:
Aim 2 of the study is to determine if the patients referred to the CHERL demonstrate health behavior improvements.

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Holtrop, PhD, Principal Investigator — Michigan State University
Locations (3):
- United States (3):
  - Genesys Health System, Flint, Michigan
  - MCRC, Grand Rapids, Michigan
  - UP Health Education Corporation, Marquette, Michigan